CLINICAL TRIAL: NCT06750419
Title: A Confirmatory, Open-label, Single-arm, Multi-centre Study to Evaluate Safety, Tolerability and Diagnostic Performance of 89Zirconium-labelled Girentuximab (89Zr-TLX250) to Non-invasively Detect Clear Cell Renal Cell Carcinoma (ccRCC) by Positron Emission Tomography/Computed Tomography (PET/CT) Imaging in Chinese Patients With Indeterminate Renal Masses (ZIRCON-CP Study)
Brief Title: 89Zr-TLX250 for PET/CT Imaging of ccRCC - ZIRCON-CP Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TLX250CDx-CP-002
Record Dates: First submitted 2024-11-26; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: 89Zr-DFO-girentuximab; 89Zr-girentuximab; 89Zr-DFO-TFP-GTX; Clear Cell Renal Cell Carcinoma (ccRCC); Indeterminate Renal Mass (IRM); ZIRCON-CP study; 89Zirconium-labelled girentuximab; 89Zr-TLX250
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm receiving the IP (Experimental): Approximately 82 evaluable adult patients will be recruited from approximately 8 renal cancer care specialist centres with access to state-of-the-art PET/CT imaging in mainland China. The number of enrolled participants may be increased to ensure sufficient confidence in measuring sensitivity and specificity of 89Zr-TLX250 PET/CT imaging.
  Following pre-screen morphological imaging to confirm evidence of IRM (to occur within 90 days of study enrolment), participants will attend a screening visit within 30 days of study enrolment, at which time baseline examinations will be undertaken.
  On Day 0, all successfully screened participants will undergo a slow IV administration of 89Zr- TLX250, at the nuclear medicine service of the respective study site. For all subjects, a PET/CT scan of the abdomen will occur on visit Day 5 (±2 days post administration [p.a.]) with nephrectomy to be performed any time after the PET/CT imaging visit, but no later than 90 days p.a. 89Zr-TLX250.
  Interventions: Drug: 89Zr-TLX250 PET/CT

INTERVENTIONS:
Drug: 89Zr-TLX250 PET/CT — 89Zr-TLX250, is a chimeric monoclonal antibody (INN name: girentuximab) with specificity for the CAIX (carbonic anhydrase 9) antigen, radiolabelled with the positron emitting radiometal zirconium- 89. Girentuximab has a CAS number of 916138-87-9. The chemical formula, without the 89Zr and the desferrioxamine, is C6460H1006N1718O2018S48 with a molecular mass of 146.5 kg/mol.
  89Zr-TLX250 is formulated as a solution for IV administration in glass vials at the nominal dosage strength of 37 MBq (±10%) for single IV use. The mass dose of 89Zr-TLX250 to be used in this Phase 3 study will be 10 mg, labelled with 37 MBq (±10%) 89Zr per dose.
  Other Names: 89Zr-DFO-girentuximab; 89Zr-girentuximab; 89Zr-DFO-TFP-GTX; 89Zirconium-labelled girentuximab

SUMMARY:
89Zr-TLX250 is under clinical development as a diagnostic agent targeting clear cell renal cell carcinoma, and this Phase 3 bridging study in mainland Chinese patients is intended to support the successful ZIRCON data (ZIRCON Clinicaltrial.gov ID: NCT03849118)

DETAILED DESCRIPTION:
This will be a confirmatory, prospective, open-label, single-arm, multi-centre study in a Chinese patient population. The study is designed to evaluate the safety, tolerability, sensitivity and specificity of 89Zr-TLX250 Positron Emission Tomography/Computed Tomography (PET/CT) imaging to non-invasively detect Clear Cell Renal Cell Carcinoma (ccRCC). The multi-centre study will be conducted in mainland China in adult patients with Indeterminate Renal Masses (IRM), who are scheduled for partial or total nephrectomy as part of their standard of care.

Approximately 82 evaluable adult patients will be recruited from approximately 8 renal cancer care specialist centres with access to state-of-the-art PET/CT imaging in mainland China. The number of enrolled participants may be increased to ensure sufficient confidence in measuring sensitivity and specificity of 89Zr-TLX250 PET/CT imaging.

The study involves a single administration of 37 MBq (±10%) of 89Zr-TLX250, containing a mass dose of 10 mg of girentuximab, in mainland Chinese participants (ZIRCON-CP). This is consistent with the confirmatory, prospective, multinational clinical trial ZIRCON (ClinicalTrials.gov ID: NCT03849118). This study consists of seven visits. Imaging will then be conducted 5±2 days post administration. The partial/total nephrectomy will then be performed at institutional discretion any time following the PET/CT imaging visit, but no later than 90 days post administration of 89Zr-TLX250. Histological tumour samples will be prepared and used for histological diagnosis of the renal mass (ccRCC or non-ccRCC) read by a central laboratory.

On Day 5±2 post study drug administration, an abdominal PET/CT imaging will be obtained. In patients, in which unexpected evidence for disseminated disease is observed, PET/CT imaging may be extended to complete whole body imaging(vertex of skull to toe) at the discretion of the investigator.

Image data analyses will be performed by a central imaging vendor.

For participants who were nephrectomised within 28 days post administration, the final study visit will be conducted on Day 42 (±7 days). For participants with nephrectomy between 28 and 90 days post administration, the final study visit will be performed 35 days (±7 days) after surgery.

Image data analyses will be performed by a central image core lab. Qualitative visual analysis (presence or absence of localised 89Zr-TLX250 uptake inside or in vicinity of renal lesion, as seen on contrast-enhanced CT or Magnetic Resonance Imaging [MRI]), will be used to assess test performance or 89Zr-TLX-250 PET/CT imaging to non-invasively detect ccRCC, using histological results from the central histological reference laboratory as standard of truth.

The duration of this study is expected to be about 12 months, with a follow-up of 4 months. The study duration for a single participant will be approximately between 4 - 6 months.

No interim analysis is planned for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Written and voluntarily given informed consent.
2. Mainland Chinese male or female, aged ≥ 18 years.
3. Imaging evidence of a single IRM of ≤ 7 cm in largest diameter (tumour stage cT1), on SoC imaging based on national standards, not older than 90 days on Day 0, but performed before any screening procedure.
4. Scheduled for lesion resection as part of regular diagnostic work-up within 90 days from planned IV 89Zr-TLX250 administration.
5. Negative serum pregnancy tests in female patients of childbearing potential at screening. Confirmation of negative pregnancy test result from urine within 24 hours prior to receiving investigational product.
6. Sufficient life expectancy to justify nephrectomy.
7. Consent to practise highly effective contraception until a minimum of 42 days after IV 89Zr-TLX250 administration.

Exclusion Criteria:

1. A biopsy procedure only (rather than partial or total nephrectomy) is planned for histological species delineation of IRM.
2. Renal mass known to be a metastasis of another primary tumour.
3. Active non-renal malignancy requiring therapy during the time frame of the study participation.
4. Multiple unilateral or bilateral IRM.
5. Chemotherapy, radiotherapy, targeted therapy or immunotherapy within 4 weeks prior to the planned administration of 89Zr -TLX250 or continuing adverse effects (> grade 1) from such therapy (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).
6. Planned antineoplastic therapies (for the period between IV administration of 89Zr-TLX250 and imaging).
7. Exposure to murine or chimeric antibodies within the last 5 years.
8. Previous administration of any radionuclide within 10 half-lives of the same.
9. Serious non-malignant disease (e.g. psychiatric, infectious, autoimmune or metabolic), that may interfere with the objectives of the study or with the safety or compliance of the study subject, as judged by the investigator.
10. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
11. Exposure to any experimental diagnostic or therapeutic drug within 4 weeks or 5 half-lives (whichever is longer) from the date of planned administration of 89Zr-TLX250.
12. Women who are pregnant or breastfeeding.
13. Known hypersensitivity to girentuximab or desferoxamine (DFO).
14. Renal insufficiency with glomerular filtration rate (GFR) ≤ 45 mL/min/1.73 m².
15. Vulnerable patients (e.g., being in detention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the sensitivity and specificity of qualitative assessment of PET/CT imaging with 89Zr-TLX250 to non-invasively detect ccRCC in patients with indeterminate renal masses, using histology as standard of truth | From Visit 4 till end of study. Diagnostic PET/CT scan on Day 5±2 days post 89Zr-TLX250 administration. Histological confirmation of the material from nephrectomy conducted within 90 days post 89Zr-TLX250 administration served as standard of truth
  Evaluating this outcome involved using a PET/CT machine on all patients to determine the uptake of the Zr89 radiotracer within the renal lesion, which was then compared to the histological determination of the lesion type following resection

SECONDARY OUTCOMES:
To determine the 89Zr-TLX250's test performance | Day of Imaging (Day 5±2 post- IP administration).
  Determine the Standardized Uptake Value (SUV) in detecting ccRCC from non-ccRCC in the kidney in the Chinese patient population.
To determine the 89Zr-TLX250's test performance | Day of Imaging (Day 5±2 post- IP administration), Post-Imaging study visit (Day 42±7 post- IP administration), Day of surgery (within 28 days post-IP administration) or Day of surgery (28 to 90 days post-IP administration).
  Determine the predictive values (%) of 89Zr-TLX250 PET/CT in detecting ccRCC from non-ccRCC in the kidney in the Chinese patient population.
To determine the 89Zr-TLX250's test performance | Day of Imaging (Day 5±2 post- IP administration), Post-Imaging study visit (Day 42±7 post- IP administration), Day of surgery (within 28 days post-IP administration) or Day of surgery (28 to 90 days post-IP administration).
  Evaluate the diagnostic accuracy (%) of 89Zr-TLX250 PET/CT in distinguishing ccRCC from non-ccRCC in the kidney in the Chinese patient population.
To assess the safety and tolerability of 89Zr-TLX250 | Day of IP administration (Day 0), Day of Imaging (Day 5±2 post- IP administration), Post-Imaging study visit (Day 42±7 post- IP administration), Day of surgery (within 28 days post-IP administration) or Day of surgery (28-90 days post-IP administration)
  Number of AEs, incidence of anti-drug antibody detection following use of the study drug in Chinese patients with IRM
To evaluate the impact of 89Zr-TLX250 PET/CT on clinical decision-making as a diagnostic tool | Day of Imaging (Day 5±2 post- IP administration), Post-Imaging study visit (Day 42±7 post- IP administration), Day of surgery (within 28 days post-IP administration) or Day of surgery (28 to 90 days post-IP administration).
  Proportion of participants with changes in management plans based on PET/CT scan findings versus conventional imaging following the use of 89Zr-TLX250

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Cancer Hospital, Beijing
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Union Hospital Tongji Medical College Huazhong University Of Science And Technology, Hubei
  - Zhongshan Hospital, Fudan University, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Cancer Hospital Airport Hospital, Tianjin
  - Affiliated Hospital Of Jiangnan University, Wuxi
  - Zhejiang Cancer Hospital, Zhejiang

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers as it is in line with ICH-GCP guidelines, which emphasise the protection of participant confidentiality and the integrity of the study data. Additionally, sharing of IPD is not planned to ensure compliance with regulatory requirements and to maintain the proprietary nature of the data.

REFERENCES:
- [Background] Shuch B, Pantuck AJ, Bernhard JC, Morris MA, Master V, Scott AM, van Praet C, Bailly C, Onal B, Aksoy T, Merkx R, Schuster DM, Lee ST, Pandit-Taskar N, Fan AC, Allman P, Schmidt K, Tauchmanova L, Wheatcroft M, Behrenbruch C, Hayward CRW, Mulders P. [89Zr]Zr-girentuximab for PET-CT imaging of clear-cell renal cell carcinoma: a prospective, open-label, multicentre, phase 3 trial. Lancet Oncol. 2024 Oct;25(10):1277-1287. doi: 10.1016/S1470-2045(24)00402-9. Epub 2024 Sep 10. PMID 39270701
- [Background] 2010 年第 7 版肾癌新分期的应用效果评估
- [Background] 肾包膜侵犯状况对于 肾癌临床症状及分期的意义
- [Background] ZIRDOSE. An open-label, Phase I study to assess safety, tolerability, radiation dosimetry, and imaging properties of 89Zr-labelled girentuximab (89Zr-girentuximab) for in vivo detection of clear cell renal carcinoma (CCRC) by positron emission tomography (PET) using different PET imaging methodologies. ClinicalTrials.gov: NCT03556046
- [Background] ZIRDAC-JP. Phase 1 open-label study to evaluate the safety/tolerability/radioactivity distribution of positron emission tomography (PET/CT) imaging with 89Zr-girentuximab (89Zr-TLX250) as well as to investigate its pharmacokinetics and pharmacodynamics in subjects with renal cell carcinoma including clear cell renal cell carcinoma (ZIRDAC-JP). ClinicalTrials.gov : NCT04496089
- [Background] ZIRCON. A confirmatory, prospective, open-label, multi-centre phase 3 study to evaluate diagnostic performance of 89Zirconium-labelled girentuximab(89Zr-TLX250) to non-invasively detect clear cell renal cell carcinoma (ccRCC) by positron emission tomography/CT (PET/CT) imaging in patients with indeterminate renal masses (ZIRCON study). ClinicalTrials.gov: NCT03849118
- [Background] Wang HY, Ding HJ, Chen JH, Chao CH, Lu YY, Lin WY, Kao CH. Meta-analysis of the diagnostic performance of [18F]FDG-PET and PET/CT in renal cell carcinoma. Cancer Imaging. 2012 Oct 26;12(3):464-74. doi: 10.1102/1470-7330.2012.0042. PMID 23108238
- [Background] van Asselt SJ, Oosting SF, Brouwers AH, Bongaerts AH, de Jong JR, Lub-de Hooge MN, Oude Munnink TH, Fiebrich HB, Sluiter WJ, Links TP, Walenkamp AM, de Vries EG. Everolimus Reduces (89)Zr-Bevacizumab Tumor Uptake in Patients with Neuroendocrine Tumors. J Nucl Med. 2014 Jul;55(7):1087-92. doi: 10.2967/jnumed.113.129056. Epub 2014 May 1. PMID 24790218
- [Background] US FDA Guidance for Industry: Multiple Endpoints in Clinical Trials January 2017 (draft) https://www.fda.gov/media/102657/download
- [Background] Stillebroer AB, Franssen GM, Mulders PF, Oyen WJ, van Dongen GA, Laverman P, Oosterwijk E, Boerman OC. ImmunoPET imaging of renal cell carcinoma with (124)I- and (89)Zr-labeled anti-CAIX monoclonal antibody cG250 in mice. Cancer Biother Radiopharm. 2013 Sep;28(7):510-5. doi: 10.1089/cbr.2013.1487. Epub 2013 May 22. PMID 23697926
- [Background] Stillebroer AB, Boerman OC, Desar IM, Boers-Sonderen MJ, van Herpen CM, Langenhuijsen JF, Smith-Jones PM, Oosterwijk E, Oyen WJ, Mulders PF. Phase 1 radioimmunotherapy study with lutetium 177-labeled anti-carbonic anhydrase IX monoclonal antibody girentuximab in patients with advanced renal cell carcinoma. Eur Urol. 2013 Sep;64(3):478-85. doi: 10.1016/j.eururo.2012.08.024. Epub 2012 Aug 21. PMID 22980441
- [Background] Steffens MG, Boerman OC, de Mulder PH, Oyen WJ, Buijs WC, Witjes JA, van den Broek WJ, Oosterwijk-Wakka JC, Debruyne FM, Corstens FH, Oosterwijk E. Phase I radioimmunotherapy of metastatic renal cell carcinoma with 131I-labeled chimeric monoclonal antibody G250. Clin Cancer Res. 1999 Oct;5(10 Suppl):3268s-3274s. PMID 10541374
- [Background] Steffens MG, Kranenborg MH, Boerman OC, Zegwaart-Hagemeier NE, Debruyne FM, Corstens FH, Oosterwijk E. Tumor retention of 186Re-MAG3, 111In-DTPA and 125I labeled monoclonal antibody G250 in nude mice with renal cell carcinoma xenografts. Cancer Biother Radiopharm. 1998 Apr;13(2):133-9. doi: 10.1089/cbr.1998.13.133. PMID 10850349
- [Background] Steffens MG, Boerman OC, Oosterwijk-Wakka JC, Oosterhof GO, Witjes JA, Koenders EB, Oyen WJ, Buijs WC, Debruyne FM, Corstens FH, Oosterwijk E. Targeting of renal cell carcinoma with iodine-131-labeled chimeric monoclonal antibody G250. J Clin Oncol. 1997 Apr;15(4):1529-37. doi: 10.1200/JCO.1997.15.4.1529. PMID 9193349
- [Background] Stabin MG, Sparks RB, Crowe E. OLINDA/EXM: the second-generation personal computer software for internal dose assessment in nuclear medicine. J Nucl Med. 2005 Jun;46(6):1023-7. PMID 15937315
- [Background] Snyder ME, Bach A, Kattan MW, Raj GV, Reuter VE, Russo P. Incidence of benign lesions for clinically localized renal masses smaller than 7 cm in radiological diameter: influence of sex. J Urol. 2006 Dec;176(6 Pt 1):2391-5; discussion 2395-6. doi: 10.1016/j.juro.2006.08.013. PMID 17085108
- [Background] Smith-Bindman R, Lipson J, Marcus R, Kim KP, Mahesh M, Gould R, Berrington de Gonzalez A, Miglioretti DL. Radiation dose associated with common computed tomography examinations and the associated lifetime attributable risk of cancer. Arch Intern Med. 2009 Dec 14;169(22):2078-86. doi: 10.1001/archinternmed.2009.427. PMID 20008690
- [Background] Schachter LR, Cookson MS, Chang SS, Smith JA Jr, Dietrich MS, Jayaram G, Herrell SD. Second prize: frequency of benign renal cortical tumors and histologic subtypes based on size in a contemporary series: what to tell our patients. J Endourol. 2007 Aug;21(8):819-23. doi: 10.1089/end.2006.9937. PMID 17867935
- [Background] Rizvi SN, Visser OJ, Vosjan MJ, van Lingen A, Hoekstra OS, Zijlstra JM, Huijgens PC, van Dongen GA, Lubberink M. Biodistribution, radiation dosimetry and scouting of 90Y-ibritumomab tiuxetan therapy in patients with relapsed B-cell non-Hodgkin's lymphoma using 89Zr-ibritumomab tiuxetan and PET. Eur J Nucl Med Mol Imaging. 2012 Mar;39(3):512-20. doi: 10.1007/s00259-011-2008-5. Epub 2012 Jan 5. PMID 22218876
- [Background] Oosting SF, Brouwers AH, van Es SC, Nagengast WB, Oude Munnink TH, Lub-de Hooge MN, Hollema H, de Jong JR, de Jong IJ, de Haas S, Scherer SJ, Sluiter WJ, Dierckx RA, Bongaerts AH, Gietema JA, de Vries EG. 89Zr-bevacizumab PET visualizes heterogeneous tracer accumulation in tumor lesions of renal cell carcinoma patients and differential effects of antiangiogenic treatment. J Nucl Med. 2015 Jan;56(1):63-9. doi: 10.2967/jnumed.114.144840. Epub 2014 Dec 4. PMID 25476536
- [Background] Oosterwijk E, Divgi CR, Brouwers A, Boerman OC, Larson SM, Mulders P, Old LJ. Monoclonal antibody-based therapy for renal cell carcinoma. Urol Clin North Am. 2003 Aug;30(3):623-31. doi: 10.1016/s0094-0143(03)00028-4. PMID 12953760
- [Background] Oosterwijk E, Ruiter DJ, Hoedemaeker PJ, Pauwels EK, Jonas U, Zwartendijk J, Warnaar SO. Monoclonal antibody G 250 recognizes a determinant present in renal-cell carcinoma and absent from normal kidney. Int J Cancer. 1986 Oct 15;38(4):489-94. doi: 10.1002/ijc.2910380406. PMID 2428759
- [Background] Muselaers CH, Stillebroer AB, Desar IM, Boers-Sonderen MJ, van Herpen CM, de Weijert MC, Langenhuijsen JF, Oosterwijk E, Leenders WP, Boerman OC, Mulders PF, Oyen WJ. Tyrosine kinase inhibitor sorafenib decreases 111In-girentuximab uptake in patients with clear cell renal cell carcinoma. J Nucl Med. 2014 Feb;55(2):242-7. doi: 10.2967/jnumed.113.131110. Epub 2014 Jan 6. PMID 24396030
- [Background] Muselaers CH, Boerman OC, Oosterwijk E, Langenhuijsen JF, Oyen WJ, Mulders PF. Indium-111-labeled girentuximab immunoSPECT as a diagnostic tool in clear cell renal cell carcinoma. Eur Urol. 2013 Jun;63(6):1101-6. doi: 10.1016/j.eururo.2013.02.022. Epub 2013 Feb 21. PMID 23453421
- [Background] Muselaers S, Mulders P, Oosterwijk E, Oyen W, Boerman O. Molecular imaging and carbonic anhydrase IX-targeted radioimmunotherapy in clear cell renal cell carcinoma. Immunotherapy. 2013 May;5(5):489-95. doi: 10.2217/imt.13.36. PMID 23638744
- [Background] Lowrance WT, Yee DS, Savage C, Cronin AM, O'Brien MF, Donat SM, Vickers A, Russo P. Complications after radical and partial nephrectomy as a function of age. J Urol. 2010 May;183(5):1725-30. doi: 10.1016/j.juro.2009.12.101. Epub 2010 Mar 17. PMID 20299040
- [Background] Loh A, Sgouros G, O'Donoghue JA, Deland D, Puri D, Capitelli P, Humm JL, Larson SM, Old LJ, Divgi CR. Pharmacokinetic model of iodine-131-G250 antibody in renal cell carcinoma patients. J Nucl Med. 1998 Mar;39(3):484-9. PMID 9529296
- [Background] Kutikov A, Fossett LK, Ramchandani P, Tomaszewski JE, Siegelman ES, Banner MP, Van Arsdalen KN, Wein AJ, Malkowicz SB. Incidence of benign pathologic findings at partial nephrectomy for solitary renal mass presumed to be renal cell carcinoma on preoperative imaging. Urology. 2006 Oct;68(4):737-40. doi: 10.1016/j.urology.2006.04.011. PMID 17070344
- [Background] The 2007 Recommendations of the International Commission on Radiological Protection. ICRP publication 103. Ann ICRP. 2007;37(2-4):1-332. doi: 10.1016/j.icrp.2007.10.003. PMID 18082557
- [Background] Hekman MCH, Rijpkema M, Aarntzen EH, Mulder SF, Langenhuijsen JF, Oosterwijk E, Boerman OC, Oyen WJG, Mulders PFA. Positron Emission Tomography/Computed Tomography with 89Zr-girentuximab Can Aid in Diagnostic Dilemmas of Clear Cell Renal Cell Carcinoma Suspicion. Eur Urol. 2018 Sep;74(3):257-260. doi: 10.1016/j.eururo.2018.04.026. Epub 2018 May 3. PMID 29730017
- [Background] Guo J, Ma J, Sun Y, Qin S, Ye D, Zhou F, He Z, Sheng X, Bi F, Cao D, Chen Y, Huang Y, Liang H, Liang J, Liu J, Liu W, Pan Y, Shu Y, Song X, Wang W, Wang X, Wu X, Xie X, Yao X, Yu S, Zhang Y, Zhou A; written; CSCO Renal Cell Carcinoma Committee. Chinese guidelines on the management of renal cell carcinoma (2015 edition). Ann Transl Med. 2015 Nov;3(19):279. doi: 10.3978/j.issn.2305-5839.2015.11.21. No abstract available. PMID 26697439
- [Background] Gaykema SB, Brouwers AH, Lub-de Hooge MN, Pleijhuis RG, Timmer-Bosscha H, Pot L, van Dam GM, van der Meulen SB, de Jong JR, Bart J, de Vries J, Jansen L, de Vries EG, Schroder CP. 89Zr-bevacizumab PET imaging in primary breast cancer. J Nucl Med. 2013 Jul;54(7):1014-8. doi: 10.2967/jnumed.112.117218. Epub 2013 May 7. PMID 23651946
- [Background] Divgi CR, Uzzo RG, Gatsonis C, Bartz R, Treutner S, Yu JQ, Chen D, Carrasquillo JA, Larson S, Bevan P, Russo P. Positron emission tomography/computed tomography identification of clear cell renal cell carcinoma: results from the REDECT trial. J Clin Oncol. 2013 Jan 10;31(2):187-94. doi: 10.1200/JCO.2011.41.2445. Epub 2012 Dec 3. PMID 23213092
- [Background] Divgi CR, Pandit-Taskar N, Jungbluth AA, Reuter VE, Gonen M, Ruan S, Pierre C, Nagel A, Pryma DA, Humm J, Larson SM, Old LJ, Russo P. Preoperative characterisation of clear-cell renal carcinoma using iodine-124-labelled antibody chimeric G250 (124I-cG250) and PET in patients with renal masses: a phase I trial. Lancet Oncol. 2007 Apr;8(4):304-10. doi: 10.1016/S1470-2045(07)70044-X. PMID 17395103
- [Background] Divgi CR, O'Donoghue JA, Welt S, O'Neel J, Finn R, Motzer RJ, Jungbluth A, Hoffman E, Ritter G, Larson SM, Old LJ. Phase I clinical trial with fractionated radioimmunotherapy using 131I-labeled chimeric G250 in metastatic renal cancer. J Nucl Med. 2004 Aug;45(8):1412-21. PMID 15299069
- [Background] Divgi CR, Bander NH, Scott AM, O'Donoghue JA, Sgouros G, Welt S, Finn RD, Morrissey F, Capitelli P, Williams JM, Deland D, Nakhre A, Oosterwijk E, Gulec S, Graham MC, Larson SM, Old LJ. Phase I/II radioimmunotherapy trial with iodine-131-labeled monoclonal antibody G250 in metastatic renal cell carcinoma. Clin Cancer Res. 1998 Nov;4(11):2729-39. PMID 9829736
- [Background] Dijkers EC, Oude Munnink TH, Kosterink JG, Brouwers AH, Jager PL, de Jong JR, van Dongen GA, Schroder CP, Lub-de Hooge MN, de Vries EG. Biodistribution of 89Zr-trastuzumab and PET imaging of HER2-positive lesions in patients with metastatic breast cancer. Clin Pharmacol Ther. 2010 May;87(5):586-92. doi: 10.1038/clpt.2010.12. Epub 2010 Mar 31. PMID 20357763
- [Background] Cheal SM, Punzalan B, Doran MG, Evans MJ, Osborne JR, Lewis JS, Zanzonico P, Larson SM. Pairwise comparison of 89Zr- and 124I-labeled cG250 based on positron emission tomography imaging and nonlinear immunokinetic modeling: in vivo carbonic anhydrase IX receptor binding and internalization in mouse xenografts of clear-cell renal cell carcinoma. Eur J Nucl Med Mol Imaging. 2014 May;41(5):985-94. doi: 10.1007/s00259-013-2679-1. Epub 2014 Mar 7. PMID 24604591
- [Background] Brouwers AH, Buijs WC, Mulders PF, de Mulder PH, van den Broek WJ, Mala C, Oosterwijk E, Boerman OC, Corstens FH, Oyen WJ. Radioimmunotherapy with [131I]cG250 in patients with metastasized renal cell cancer: dosimetric analysis and immunologic response. Clin Cancer Res. 2005 Oct 1;11(19 Pt 2):7178s-7186s. doi: 10.1158/1078-0432.CCR-1004-0010. PMID 16203819
- [Background] Brouwers AH, van Eerd JE, Frielink C, Oosterwijk E, Oyen WJ, Corstens FH, Boerman OC. Optimization of radioimmunotherapy of renal cell carcinoma: labeling of monoclonal antibody cG250 with 131I, 90Y, 177Lu, or 186Re. J Nucl Med. 2004 Feb;45(2):327-37. PMID 14960657
- [Background] Brouwers AH, Buijs WC, Oosterwijk E, Boerman OC, Mala C, De Mulder PH, Corstens FH, Mulders PF, Oyen WJ. Targeting of metastatic renal cell carcinoma with the chimeric monoclonal antibody G250 labeled with (131)I or (111)In: an intrapatient comparison. Clin Cancer Res. 2003 Sep 1;9(10 Pt 2):3953S-60S. PMID 14506194
- [Background] Brouwers AH, Dorr U, Lang O, Boerman OC, Oyen WJ, Steffens MG, Oosterwijk E, Mergenthaler HG, Bihl H, Corstens FH. 131 I-cG250 monoclonal antibody immunoscintigraphy versus [18 F]FDG-PET imaging in patients with metastatic renal cell carcinoma: a comparative study. Nucl Med Commun. 2002 Mar;23(3):229-36. doi: 10.1097/00006231-200203000-00005. PMID 11891480
- [Background] Borjesson PK, Jauw YW, de Bree R, Roos JC, Castelijns JA, Leemans CR, van Dongen GA, Boellaard R. Radiation dosimetry of 89Zr-labeled chimeric monoclonal antibody U36 as used for immuno-PET in head and neck cancer patients. J Nucl Med. 2009 Nov;50(11):1828-36. doi: 10.2967/jnumed.109.065862. Epub 2009 Oct 16. PMID 19837762
- [Background] Andersson M, Johansson L, Eckerman K, Mattsson S. IDAC-Dose 2.1, an internal dosimetry program for diagnostic nuclear medicine based on the ICRP adult reference voxel phantoms. EJNMMI Res. 2017 Nov 3;7(1):88. doi: 10.1186/s13550-017-0339-3. PMID 29098485
- See also: IPD registration in Chinadrugtrials as per Chinese requirements — http://www.chinadrugtrials.org.cn/